CLINICAL TRIAL: NCT06511219
Title: Evaluation of Maxillary Segmental Distalization Using Infra Zygomatic Versus Palatal Digitally Printed Skeletal Anchored Appliances
Brief Title: Maxillary Segmental Distalization Using Digitally Printed Appliances
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Elabd, teaching assistant - orthodontic department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: phd
Record Dates: First submitted 2024-06-21; First posted 2024-07-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-07

CONDITIONS: Class II Malocclusion
Keywords: class II maloccluusion, miniscrew
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Intervention Model Description: The buccal segmental distalizer will take the anchorage from infrazygomatic miniscrews (IZC).
  the palatal distalizer take anchorage from palate
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- maxillary segmental distalization using infrazygomatic digitally printed appliances (Active Comparator): maxillary segmental distalization using infrazygomatic digitally printed appliances
  Interventions: Device: maxillary segmental distalization
- maxillary segmental distalization using palatal digitally printed appliances (Active Comparator): maxillary segmental distalization using palatal digitally printed appliances
  Interventions: Device: maxillary segmental distalization

INTERVENTIONS:
Device: maxillary segmental distalization — maxillary segmental distalization using skeletal anchored digitally printed appliances

SUMMARY:
Evaluation of Maxillary Segmental Distalization Using Infrazygomatic versus Palatal Digitally Printed Skeletal Anchored Appliances.

DETAILED DESCRIPTION:
Ethical approval All selected patients will be informed about the aims and characteristics of the study, the potential risks and benefits and the option of withdrawing from it whenever they desire. Then all patients will sign the informed consent document. All patients will be informed about the results after finishing. All selected patients' personal data and details will be held and handled confidentially and privately in the orthodontic department, faculty of dentistry, Mansoura university.

Trial design

Patients will be randomly allocated into two groups as follow:

1. First group: Buccal segmental digitally printed maxillary distalizer (infrazygomatic mini-implant IZC).
2. Second group: palatal segmental digitally printed maxillary distalizer.

The buccal segmental distalizer will take the anchorage from infrazygomatic miniscrews.

The distalizer will be composed of digitally printed metal shell which is bonded to the palatal surface of the whole posterior segment.

Transpalatal arm will connect the two sides to avoid buccal tipping during distalization.

The distalization will be done by placing chain elastics from the miniscrews to the hook present in the mesial aspect of the appliance.

The palatal segmental distalizer will take anchorage from miniscrews placed in the anterior palate.

The appliance will be bonded to the palatal surface of the posterior segment and containing two anterior and two posterior hooks.

The distalization will be performed by using chain elastics between the anterior and posterior hooks.

Force: 300-350 gram per side which will be measured using force gauge.

A follow-up session will be scheduled every 3weeks, and the appliance will be removed in both groups after the patient reach a Class I relationship. For each patient, two lateral cephalograms will be obtained: one preoperatively and another after completion of distalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients age (13- 18) years.
* Full permanent dentition except third molar.
* Class II malocclusion with at least an end-on Class II molar relationship bilaterally.
* normal or short lower facial height.

Exclusion Criteria:

* Systemic conditions that may interfere with the treatment.
* Bad habits that might jeopardize the appliance.
* Transverse discrepancy.
* Previous orthodontic treatment.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Maxillary Segmental Distalization Using Infrazygomatic versus Palatal Digitally Printed Skeletal Anchored Appliances. | 10 months
  this study includes 40 patients with class II molar and canine relation the study aimes to investigate the effect of the skeletal anchored digitally printed distalizers on the distal movement of the maxillary posterior segment in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No